CLINICAL TRIAL: NCT00960258
Title: Phase I, Uncontrolled, Open-label, Non-randomized Study to Investigate Pharmacokinetics and Safety of BAY73-4506 in Asian (Japanese) Patients With Advanced, Refractory Solid Tumors
Brief Title: Phase I Study to Investigate Pharmacokinetics and Safety of BAY73-4506 in Asian (Japanese) Patients With Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13172
Record Dates: First submitted 2009-07-03; First posted 2009-08-17 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Tumors
Keywords: Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Regorafenib (BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506) — The patients will be treated on Day 1 of the first week followed by 6 days off treatment (Cycle 0, single dosing period). After Cycle 0, the patients will be treated with BAY 73-4506 (160 mg once daily orally, 21 days on/ 7 days off schedule). Dose level : 160 mgDose level-1: 120 mgDose level-2: 60 mg

SUMMARY:
This study is to define the pharmacokinetics and to evaluate the safety of BAY73-4506, 160 mg once daily administered orally as a single agent in Japanese patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese patients >/= 18 years
* Histologically or cytologically confirmed solid tumors
* ECOG-PS 0 - 1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Uncontrolled hypertension
* Patients with severe renal impairment or on dialysis
* Patients with seizure disorder requiring anticonvulsant medication
* Known or suspected allergy to the investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2013-11-11 (Actual)

PRIMARY OUTCOMES:
Grade 4 neutropenia for >/= 7 days, febrile neutropenia with Grade 4 neutropenia, Grade 4 thrombocytopenia, Grade 3 or 4 non-hematologic toxicity, hypertension and skin toxicity of Grade 3 or 4 which are not manageable and pharmacokinetics | After 5 weeks (after Cycle 1).

SECONDARY OUTCOMES:
Biomarker | At screening
Response rate | Every 8 weeks for the first 6 cycles. After Cycle 6, every 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Japan (4):
  - Kashiwa-shi, Chiba
  - Hidaka, Saitama
  - Chuo-ku, Tokyo
  - Mitaka, Tokyo